CLINICAL TRIAL: NCT04608656
Title: Livestock Programming for Nutritional Improvements in Pregnant, Lactating Mothers and Children Under Five Years of Age in Marsabit County, Kenya
Brief Title: Livestock for Health Project
Acronym: L4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Food and Agriculture Organization of the United Nations (Unknown); UNICEF (Other)
Responsible Party: Principal Investigator, Thumbi Mwangi, Research Associate Professor, Washington State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: KEMRI/SERU/CGHR/02-09/3755
Record Dates: First submitted 2020-10-07; First posted 2020-10-29 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Malnutrition
Keywords: Children under five years; Pregnant and Lactating women; Livestock feeds; Nutrition counselling; Undernutrition; Pastoralism; Kenya
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: The study households will be assigned one of three study arms:
  i) Intervention arm 1: Livestock feed only.
  Households in villages assigned to intervention arm 1 will receive a pre-defined amount of livestock feed to maintain two tropical livestock units for a total of 60 days during the dry season (when animals would be moved away in search of pastures).
  ii) Intervention arm 2: 1.Provision of Livestock feed, 2. Nutritional counselling
  Households recruited into intervention arm two will receive livestock feeds and will be enrolled in a nutritional education and counselling program.
  iii) Control arm
  The households recruited under this arm will receive none of the two study interventions. These households will receive identical assessment and data collection like other study households in the study.
Who Masked: Participant, Investigator
Masking Description: Data collection enumerators will not be aware which intervention arm the households belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm 1: Livestock feed only (Experimental): Households in villages assigned to intervention arm 1 will receive a pre-defined amount of feed to maintain two tropical livestock units for a total of 60 days during the dry season (when animals would be moved away in search of pastures).
  Interventions: Other: Provision of livestock feeds
- Intervention arm 2: 1. Provision of Livestock feeds, 2. Nutrition counselling (Experimental): Households recruited into intervention arm two will receive livestock feeds similar to intervention arm 1 and will be enrolled in a nutritional education and counselling program through Infant and Young Child Nutrition (IYCF) feeding program and household food utilization. The IYCF program through the Baby Friendly Community Initiative (BFCI) will include the promotion of exclusive breastfeeding in the first six months, continued breastfeeding up to the age of two years, adequate complementary feeding, hygiene promotion and the uptake of child health services including immunization, treatment of illness, moderate and severe acute malnutrition and micro-nutrient supplementation.
  Interventions: Other: Provision of livestock feeds; Other: Nutrition counselling
- Control arm (No Intervention): The households recruited under this arm will receive none of the two study interventions. These households will receive identical assessment and data collection like other study households in the study. Their access to support through other interventions will be monitored. Households within the control arm will receive nutritional counselling and education given outside of the project. This is mainly at health facilities when mothers present for antenatal care or visit health facilities seeking healthcare. On some occasions in places where community health volunteers are present, nutritional counselling and education may be provided at the community level. The study instruments have been designed to collect information at the household level if such nutritional counselling and education has been provided.

INTERVENTIONS:
Other: Provision of livestock feeds — Households will receive livestock feeds (ranch cubes) for the select lactating animals during the dry season
  Arms: Intervention arm 1: Livestock feed only; Intervention arm 2: 1. Provision of Livestock feeds, 2. Nutrition counselling
Other: Nutrition counselling — Households will receive livestock feeds (ranch cubes) for the select lactating animals and will also be enrolled in to a nutrition counselling programme
  Arms: Intervention arm 2: 1. Provision of Livestock feeds, 2. Nutrition counselling

SUMMARY:
Children 5 years and below, and pregnant/lactating women in pastoralist communities suffer a high burden of acute malnutrition. Improving the health and productivity of animals can reduce the risk malnutrition during the dry periods. The aim of this study is to assess how providing livestock with feeds during critical dry periods can improve household milk availability, consumption and risk of malnutrition in pregnant and lactating mothers, and children 5 years and below.

The study will be a cluster randomized control trial conducted in Marsabit County and will involve a total of 1800 households that own livestock and have children 5 years and below. The households will be divided into three groups and each group will have a total of 600 households. Group one, will receive livestock feed enough to maintain 2-3 milking animals during the critical dry period. The second group will receive similar livestock feed but will also receive education and counselling on human nutrition. The third group will be the control arm and will not receive any of the two interventions.

The study will aim to estimate how these interventions impact stunting and underweight in children and weight gain for pregnant women by collecting data on middle upper arm circumference, height, weight, and weight-gain during pregnancy every three months in a year. In addition, data on food consumption patterns such as number of meals taken, type/diversity of foods consumed including animal source foods, frequency of times and quantity of specific foods consumed) on at least 6-weekly basis will be collected. To further understand this problem the investigators will collect human illness data including on fever, diarrhoea, and respiratory syndromes among study participants during the regular visits. Socio-economic data including household demographics, incomes, expenditures, asset accumulation, gender roles, and workload and time allocation will be collected quarterly. Biological samples will be collected (venous blood and mother's milk) at recruitment, six months and 12 months. Screening for infections such as brucellosis, micronutrient and mycotoxin analysis will be conducted on the biological samples in order account for infections or conditions that could have an impact on nutritional status of study participants. The study will also assess which of the interventions provide value for money given that resources are scarce.

DETAILED DESCRIPTION:
Background: In households heavily dependent on livestock, declining availability of forage is associated with decreased consumption of animal source foods such as milk and meat, and consequently decline in child nutritional status. Populations living in Kenya's Arid and Semi-Arid Lands(ASALs) are predominantly pastoral, heavily dependent on livestock and practice seasonal mobility to access livestock pasture and water. Livestock interventions that maintain or improve health and productivity of animals have been postulated as important for reducing the risk of malnutrition during critical drought periods.

Objectives: Here the investigators implement a cluster randomized control study trial to determine the effect of providing livestock feed, livestock feed and nutritional education and counselling during critical dry periods on household milk availability and consumption, and the risk of malnutrition in pregnant and lactating mothers, and children 5 years and below.

Methods: A total of 1800 households owning livestock and with children 3 years and below in Marsabit County will be enrolled into three equal groups (arms) of 600 households each. Each household and participant will be followed for 18 months. Households in Arm 1 will receive livestock feed enough to maintain 2-3 milking animals during the critical dry period. Arm 2 will receive similar livestock feed and human nutritional education and counselling. Arm 3 (control arm) will not have any of the two interventions. Primary outcome measures will be child anthropometric indicators (height-for-age, weight-for-age and middle upper arm circumference) and maternal anthropometric measures (middle upper arm circumference, height, weight, weight-gain during pregnancy) collected quarterly. Data on a 24-hour recall of diet (number of meals taken, type/diversity of foods consumed including animal source foods, frequency of times and quantity of specific foods consumed) will be collected every 6 weeks. To control for additional factors that would influence nutritional status, the investigators will collect human health syndromic data (fever, diarrhoea, respiratory syndromes) and livestock health data every six weeks and socio-economic data quarterly including household demographics, incomes, expenditures, asset accumulation, gender roles, workload and time allocation. To control for exposure to infections such as brucellosis in humans and animals and for micronutrient and mycotoxin analysis, biological samples (venous blood of mother and child), animal biological samples (blood and milk) and household drinking water will be collected at recruitment, 6 months and at 12 months. The study will test the cost-effectiveness of livestock interventions and nutritional counselling in prevention of malnutrition and its health consequences, compared to treatment of malnutrition. Cost data associated with each study arm will be tracked to provide estimates of resources required to scale up for implementation. Results from this study will form the basis for monitoring efficiency and effectiveness of interventions aimed at reducing seasonal spikes in levels of acute malnutrition in children under five years and pregnant and lactating women in pastoralist communities.

Study duration: Each study household and participant is followed for a period of 24 months from the time of enrolment into the study.

ELIGIBILITY:
Inclusion Criteria:

* Household inclusion criteria

Only households meeting the following study criteria will be recruited:

* Presence of a mother (lactating or non-lactating) and child 3 years and below
* Ownership of livestock with 1-6 tropical livestock units
* Household consent to participate in the study o Including willingness to have 1-2 tropical livestock units (1-2 cattle or camel, 10-20 sheep/ goats) at household

Exclusion Criteria:

* Households excluded in the study will have the following criteria:

  * Households that do not consent to participate in the study
  * Households unwilling to adhere to the study protocol including feeding instructions and retaining the study animals at the household for milk access

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1734 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Household milk yield (litres/week) | 24 months
  Compare the household milk yield in liters per week between the three study arms.
  Average amount of milk produced per week by species (cattle, camels, goats and sheep)compare mean change in household average milk yield (litres/week) over study time by the intervention and control study arms.
Milk consumption (amount and frequency) by children < 5 years and pregnant and lactating women | 24 months
  Compare the average daily milk intake for mothers and children participating in the study between the three study arms.
Undernutrition (wasting, stunting and underweight) | 24 months
  Determine the levels and trends of undernutrition(wasting, stunting and underweight) among children < 5 years and pregnant and lactating women
Cost-effectiveness ratio of (changes in total cost of interventions by arm )/(Changes in acute malnutrition (WHZ) by arm) | 24 months
  Determine if providing livestock feed, livestock feed and nutritional counselling is a cost-effective way of preventing acute malnutrition in children < 5 years and mothers.
  A cost-effective analysis will be used to complete an economic assessment of the costs of malnutrition and treatment of malnutrition in the absence of livestock feed intervention, and livestock feed and nutritional counseling intervention. Costs will be quantified using intervention, treatment and economic data (including market prices and household sales) collected over the period of the study.
  The cost-effectiveness analysis will be conducted in two stages;
  1. based on the changes in the acute malnutrition ($/WHZ) between the intervention arms and control arm, and
  2. using standardized measure encompassing both morbidity and mortality associated with malnutrition - cost per quality-adjusted life years (QALYs) gained or disability-adjusted life years (DALYs) averted .

CONTACTS AND LOCATIONS:
Overall Officials: Thumbi Mwangi, PhD, Principal Investigator — Washington State University, Paul G Allen School for Global Animal Health; Josphat M Muema, PhD(c), Study Director — Washington State University - Global Health Kenya; Mutono Nyamai, PhD(c), Study Director — Washington State University - Global Health Kenya; Guy Palmer, PhD, Study Chair — Washington State University, Paul G Allen School for Global Animal Health
Locations (1):
- Washington State University, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
A repository/database with all IPD that underlie results in all publications generated from the study will be developed
Supporting Information: Study Protocol, SAP
Time Frame: When the study articles have been published
Access Criteria: On request

REFERENCES:
- [Derived] Thumbi SM, Muema J, Mutono N, Njuguna J, Jost C, Boyd E, Tewoldeberhan D, Mutua I, Gacharamu G, Wambua F, Allport R, Olesambu E, Osman AM, Souza D, Kimani I, Oyugi J, Bukania Z, Oboge H, Palmer GH, Yoder J. The Livestock for Health Study: A Field Trial on Livestock Interventions to Prevent Acute Malnutrition Among Women and Children in Pastoralist Communities in Northern Kenya. Food Nutr Bull. 2023 Dec;44(2_suppl):S119-S123. doi: 10.1177/03795721231195427. PMID 37850922